CLINICAL TRIAL: NCT06834802
Title: 3D Analysis of Soft Tissue Healing After Immediate Implant Placement in Molar Sites Using PRF Vs HAM: A Randomized Controlled Clinical Study in Molar Sites Using PRF Vs HAM: A Randomized Controlled Clinical Study
Brief Title: 3D Analysis of Soft Tissue Healing After Immediate Implant Placement Using PRF Vs HAM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3D soft tissue assessment
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Badly Broken Maxillary Premolars Indicated for Extraction; Badly Broken Down Vital Teeth
Keywords: jumping gap; immediate implant placemnet; soft tissue around implant; soft tissue healing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of outcome assessors and participants will be achieved as the different outcomes will be assessed for all groups by assessors other than the researchers doing the procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Grafting with PRF (Active Comparator): immediate implant will be placed and PRF membrane will be placed into the soft tissue. The PRF plug will be maintained in place with approximating sutures using 5-0 resorbable suture material.
  Interventions: Procedure: PRF
- Grafting using Human amniotic membrane (HAM) (Active Comparator): immediate implant placement will be done and The HAM plug will be placed into the soft tissue.
  Interventions: Procedure: Human amniotic membrane
- No Grafting (Active Comparator): Immediate implant placement will be done and with no soft tissue grafting
  Interventions: Procedure: No grafting

INTERVENTIONS:
Procedure: PRF — PRF membrane will be used for soft tissue grafting around implant
  Arms: Grafting with PRF
Procedure: Human amniotic membrane — Human amniotic membrane will be used for soft tissue grafting around implan
  Arms: Grafting using Human amniotic membrane (HAM)
Procedure: No grafting — No soft tissue grafting around implant
  Arms: No Grafting

SUMMARY:
Statement of the problem: Soft tissue healing following immediate implant placement is one of the major factors that affect implant restoration, function & success.

Aim: The aim of this study is to compare the effect of using HAM (Human amniotic membrane) and platelet rich fibrin (PRF) in soft tissue healing with immediate implant placement in the molar region.

DETAILED DESCRIPTION:
Aim: The aim of this study is to compare the effect of using HAM (Human amniotic membrane) and platelet rich fibrin (PRF) in soft tissue healing with immediate implant placement in the molar region.

Materials and Methods: This parallel arm, randomized controlled clinical trial will involve systemically free patients with remaining roots or badly decayed teeth in molar sites region requiring implant placement. They will be randomly allocated to three equal groups. Group A (test group, n=12) will receive immediate implants (grafting with PRF), group B (test group, n=12) will receive immediate implants (grafting with HAM) and group c (test group, n=12) will receive immediate implants (no grafting). After implant placement, soft tissue healing (1ry outcome) and postoperative pain (2nd outcome) will be assessed. The parameters will be assessed at baseline, every day for the first week, day after day second week, once in third and fourth week. Postoperative pain and swelling will be recorded daily by the patient for the 1st two weeks post surgically. Postoperative medication will be prescribed to the patient and postoperative instructions will be explained in detail. Follow-up will be performed to assess the parameters and to ensure performing proper oral hygiene. Data collected will be tabulated and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 18 years old, with non-restorable first and second molars.
2. Minimum remaining alveolar height of four to six millimeters distance from the apex of the socket to the floor of maxillary sinus for maxillary teeth and minimum remaining alveolar height of six millimeters distance from the apex of the socket to the inferior alveolar nerve for mandibular teeth.
3. Minimum alveolar Bucco-palatal dimension of 7 mm.

Exclusion Criteria:

1. Patients with known systemic diseases which can affect normal bone formation or blood coagulation.
2. Patients who are smokers.
3. Presence of signs of active infection or pus formation.
4. Absence or loss of buccal wall prior to implant placement.
5. Bad oral hygiene

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Soft tissue healing | Baseline, every day for the first week, day after day second week, once in third and fourth week
  Surface area/intraoral scanner

SECONDARY OUTCOMES:
post operative pain | Baseline, every day for the first week, day after day second week, once in third and fourth week
  Visual analog scale: numerical scale in which 0 is no pain and 10 is maximum pain

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of oral and dental medicine , Suez university, Cairo, Cairo Governorate, Egypt